CLINICAL TRIAL: NCT06157697
Title: Social Transfers for Exclusive Breastfeeding in São Paulo, Brazil
Brief Title: Social Transfers for Exclusive Breastfeeding in Brazil
Acronym: STEBB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Tropical & Public Health Institute (Other)
Collaborators: University of Sao Paulo (Other); University of Basel (Other); Swiss National Science Foundation (Other); Federal University of São Paulo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: steb2
Record Dates: First submitted 2023-11-27; First posted 2023-12-06 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2024-09

CONDITIONS: Breast Feeding, Exclusive; Breastfeeding; Development, Child; Development, Infant
Keywords: exclusive breastfeeding; child development; social transfer
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control Group (No Intervention): Only educational materials focused on the benefits of exclusive breastfeeding and the current international recommendations are provided.
- Intervention Group 1 - Non-Conditional Social Transfer (Experimental): Educational materials focused on the benefits of exclusive breastfeeding and the current international recommendations are provided. At the baseline visit, participants are told that at the 6-month visit, they will receive a gift of their choice - which is meant to show our appreciation and support for their efforts in breastfeeding.
  Intervention: Behavioral: Social Transfer
  Interventions: Behavioral: Social Transfer
- Intervention Group 2 - Conditional Social Transfer (Experimental): Educational materials focused on the benefits of exclusive breastfeeding and the current international recommendations are provided. At the baseline visit, participants are told that at the 6-month visit, they will receive a gift of their choice if they are still exclusively breastfeeding.
  Intervention: Behavioral: Social Transfer
  Interventions: Behavioral: Social Transfer

INTERVENTIONS:
Behavioral: Social Transfer — Social transfers are defined as a cash or in-kind transfer. Based on previous social transfer programs in Brazil, we will offer gift packages for mothers at 6 months. The options include: diapers, hygiene products, child developmental toys, transport vouchers, or a combination of these.
  Arms: Intervention Group 1 - Non-Conditional Social Transfer; Intervention Group 2 - Conditional Social Transfer

SUMMARY:
The goal of this study is to assess the effectiveness of social transfers on exclusive breastfeeding rates in São Paulo, Brazil. The main research questions are:

1. Are social transfers effective at increasing exclusive breastfeeding rates
2. Are social transfers effective in prolonging the duration of exclusive breastfeeding
3. Are social transfers effective in prolonging the duration of complementary breastfeeding
4. What are the long-term impacts of social transfers for breastfeeding on child health and development

Participants will be randomly assigned to one of three groups: 1) control, no social transfer 2) non-conditional social transfer at 6-months postpartum, and 3) conditional social transfer at six months postpartum; conditional upon the mothers exclusive breastfeeding status.

All participants receive education about the benefits of exclusive breastfeeding and current international recommendations.

Researchers will compare the intervention groups to the control group to see if social transfers are effective at increasing exclusive breastfeeding rates at six months postpartum.

ELIGIBILITY:
Inclusion Criteria:

* Gave birth in the last 72 hours
* Exclusively breastfeeding at time of recruitment and intend to continue to exclusively breastfeed
* Part of or eligible Bolsa Familia or on the Bolsa Familia list (CAD Unico)
* Lives in São Paulo
* No illnesses that contraindicates breastfeeding
* Had a healthy singleton infant of 37 weeks or more gestation with a birth weight of at least 2500 grams
* Agrees to participate and sign an informed consent; if under age (12-17 years), a legal representative will also have to agree to sign the informed consent

Exclusion Criteria:

* Plans to move permanently outside study area
* Has a medical, intellectual or psychological disability
* Contraindication for breastfeeding
* Preterm births
* Children born with < 2500 grams

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-03-06 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Exclusive Breastfeeding | 6 months postpartum
  The proportion of women exclusively breastfeeding at 6-months postpartum will be assessed using a questionnaire. Exclusive breastfeeding is defined as receipt of only human milk - which is consistent with the World Health Organization guidelines. At six months postpartum, mothers are asked if they are still currently breastfeeding. If they answer yes, a follow-up question on if they provided any other liquids, solids, or supplements to their child to determine the exclusive breastfeeding status.
Duration of Exclusive Breastfeeding | 6 months postpartum
  The duration of exclusive breastfeeding will be assessed using a questionnaire. Exclusive breastfeeding is defined as receipt of only human milk - which is consistent with the World Health Organization guidelines. At six months postpartum, mothers are asked if they are still currently breastfeeding. If they answer yes, a follow-up question on if they provided any other liquids, solids, or supplements to their child to determine the exclusive breastfeeding status.

SECONDARY OUTCOMES:
Child Health Outcomes | 1 month, 6 months, 1 year, 2 years
  We will assess the child's health outcomes by using a questionnaire. The questionnaire will ask a range of yes or no questions about disease/illness history, hospitalizations, and other health events.
Early Childhood Development | 1 year, 2 years
  When the child is two years of age, a comprehensive end line assessment will be conducted to evaluate early childhood development indicators (e.g. The Global Scale for Early Development (GSED). This indicator will be normalized to a mean of 0 and a standard deviation of 1 to facilitate interpretation of estimated group differences.
Prevalence of Complementary Breastfeeding | 6 months, 1 year, 2 years
  The proportion of women complementary breastfeeding at 1-year, and 2-years postpartum will be assessed using a questionnaire. Complementary breastfeeding is defined as receipt of human milk in combination with complementary foods and liquid. At each time point postpartum, mothers are asked if they are still currently breastfeeding. If they answer yes, a follow-up question on if they provided any other liquids, solids, or supplements to their child to determine the complementary breastfeeding status.
Duration of Complementary Breastfeeding | 6 months, 1 year, 2 years
  The duration of complementary breastfeeding at 1-year, and 2-years postpartum will be assessed using a questionnaire. Complementary breastfeeding is defined as receipt of human milk in combination with complementary foods and liquid. At each time point postpartum, mothers are asked if they are still currently breastfeeding. If they answer yes, a follow-up question on if they provided any other liquids, solids, or supplements to their child to determine the complementary breastfeeding status.

CONTACTS AND LOCATIONS:
Overall Officials: Jordyn Wallenborn, Principal Investigator — Swiss Tropical & Public Health Institute
Locations (2):
- Brazil (2):
  - University of Sao Paulo, São Paulo, Butantã
  - Federal University of São Paulo, São Paulo

REFERENCES:
- [Derived] Khoury S, Brentani A, Brentani H, Fiamoncini J, Francisco R, Onofre AC, Rodrigues Henrique SE, Fink G, Wallenborn J. Social Transfers for Exclusive Breastfeeding in Brazil: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 Sep 24;14:e75796. doi: 10.2196/75796. PMID 40991943